CLINICAL TRIAL: NCT05294991
Title: Consumer-Based Meditation App, Calm, for Treatment of Sleep Disturbance in Hematological Cancer Patients
Brief Title: Wellness App for Sleep Disturbance in Hematological Cancer Patients
Acronym: Heme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Arizona State University (Other); Laboratory Corporation of America (Industry); Wake Forest University Health Sciences (Other); Calm.com, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CTMS# 22-0116; R01CA262041 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Sleep Disturbance; Anxiety; Depression; Inflammation; Fatigue
MeSH Terms: conditions — Neoplasms; Parasomnias; Anxiety Disorders; Depression; Inflammation; Fatigue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness app intervention #1 (Experimental): Participants assigned to this group will be asked to engage with the app a minimum of 10 minutes per day (70 minutes per week), at any time of day they choose for at 8-week period. There is a recommended program to follow for the 8-week period, but participants are also welcome to engage with other features and content within the app.
  Interventions: Behavioral: Wellness app intervention #1
- Wellness app intervention #2 (Active Comparator): Participants assigned to this group will be asked to engage with the app a minimum of 10 minutes per day (70 minutes per week), at any time of day they choose for at 8-week period. There is a recommended program to follow for the 8-week period, but participants are also welcome to engage with other features and content within the app.
  Interventions: Behavioral: Wellness app intervention #2

INTERVENTIONS:
Behavioral: Wellness app intervention #1 — This is the active intervention group.
  Arms: Wellness app intervention #1
Behavioral: Wellness app intervention #2 — This is the active comparator/control group.
  Arms: Wellness app intervention #2

SUMMARY:
In a randomized controlled trial (RCT), the investigators will recruit participants to an 8-week "app-based wellness" intervention, followed by a 12-week follow-up period. The investigators will recruit a total of 276 self-declared Chronic Hematological Cancer (CHC) patients who (representative of age, race/ethnicity, and gender) will be on stable CHC pharmacologic therapy (if any), self-identify as sleep disturbed (>5 on Pittsburgh Sleep Quality Index), do not have a sleep disorder diagnosis, do not take sleep medication/supplements >3 times per week, and are not currently practicing regular meditation.

Aim 1: Test the efficacy of two app-based wellness programs (10 minutes per day) on the primary outcome of self reported sleep disturbance (Insomnia Severity Index (primary) and PROMIS Sleep Disturbance (secondary)) and secondary sleep outcomes including sleep impairment (PROMIS Sleep Impairment Scale) and sleep efficiency measured via sleep diaries and actigraphy.

Aim 2: Test the efficacy of two app-based wellness programs (10 minutes per day) on inflammatory markers (i.e., TNF-a, IL-6, IL-8, CRP), fatigue, and emotional distress (i.e., anxiety, depressive symptoms measured with PROMIS®).

Aim 3: Explore the sustained effects (i.e., 20 weeks from baseline) of two app-based wellness programs (10 minutes per day) in CHC patients.

DETAILED DESCRIPTION:
Background:

Hematological cancers account for 11% of all cancer diagnoses in the US. Chronic hematological cancer (CHC) patients are characterized by long term and high symptom burden. Up to 65% of CHC patients report chronic sleep disturbances (e.g., difficulty falling asleep, difficulty staying asleep, nonrestorative sleep, insomnia) that are highly correlated with poorer cognitive and physical functioning, increases in fatigue and emotional distress, and heightened levels of specific inflammatory markers (TNF-a, IL-6, IL-8, CRP) that negatively impact quality of life. Sleep interventions have been tested in solid tumor patients, but no research has examined sleep interventions specifically for CHC patients. Medications are commonly prescribed but often come with side effects and risk for long-term dependence. Cognitive behavioral therapy for insomnia (CBT-I) is the most studied and first line of therapy for treating sleep disturbances in cancer patients, but CBT-I is time-consuming, resource-intensive, and not easily accessible for all cancer patients. There is a need for long-term, accessible, non-pharmacologic interventions targeting sleep in CHC patients.

RCTs have shown meditation and mindfulness-based interventions lead to improvements in sleep disturbance among breast cancer patients, but this research has not been extended to CHCs. Meditation has potential as a non-pharmacologic strategy to reduce sleep disturbance in CHC patients without the time and expertise limitations of CBT-I and side effect risks from medication. In person meditation, however, is still inaccessible long term due to potential fatigue, pain, transportation, and scheduling difficulties.

Smartphone apps have attracted considerable interest from cancer patients as an easily accessible and empowering way to self-manage health. Existing research using apps has focused on short term psychological measures (e.g., distress, cancer-related distress, anxiety, etc.) or cancer-specific biological changes as outcomes and not sleep disturbance, in solid tumor survivors with minimal residual disease (e.g., breast cancer post-treatment), or those with short survival (e.g., metastatic solid tumor patients). The unique, long-lasting disease course of CHC patients and high chronic symptom burden warrants distinct interventions from resolved solid tumor patients. CHC patients with sleep disturbance have no options for easily accessible and evidence-based treatments for sleep disturbances. The investigators propose to test the effects of two app-based wellness programs (10 minutes per day) on sleep disturbance in CHC patients.

Study Timeline:

This study is expected to last 5 years with enrollment beginning in January 2023. The investigators aim to enroll 276 CHC patients.

Objectives:

Objective #1: Test the efficacy of two app-based wellness programs (10 minutes per day) on the primary outcome of self-reported sleep disturbance (Insomnia Severity Index (primary) and PROMIS Sleep Disturbance (secondary) and additional secondary sleep outcomes including sleep impairment (PROMIS Sleep Impairment Scale) and sleep efficiency measured via sleep diaries and actigraphy.

Objective #2: Test the efficacy of two app-based wellness programs (10 minutes per day) on inflammatory markers (i.e., TNF-a, IL-6, IL-8, CRP), fatigue, and emotional distress (i.e., anxiety, depressive symptoms measured with PROMIS®).

Objective #3: Explore the sustained effects (i.e., 20 weeks from baseline) of two app-based wellness programs (10 minutes per day) on in CHC patients.

Recruitment:

The investigators aim to recruit 276 CHC patients nationally.

Study Procedures:

All study procedures are remote and have been approved by an institutional review board. Interested patients will complete an online eligibility survey via RedCap. Eligible participants will be sent an email notifying them of their eligibility, asked to review a video-based overview of the study. If interested in participating, participants will be invited to electronically sign the informed consent via RedCap.

Once the consent is signed, participants will receive information on how to provide a blood sample at a local lab, how to choose a size for their sleep device, and sign up for a 30-minute virtual visit with a research assistant. Once participants receive their sleep device in the mail, they will meet with a research assistant via video conference to review the study procedures and activate their sleep device. After the video conference, participants will be sent an online link to complete the baseline survey. Then, for 7 days (baseline week), participants will be asked to wear a sleep device continuously and complete an online sleep diary each morning upon waking. At the end of the baseline week, participants will receive compensation and will then be randomized to download one of two wellness apps.

During the 8-week intervention period, participants will be asked to wear the sleep device continuously and complete an online sleep diary each morning. They will also be asked to engage with their assigned wellness app each day for at least 10 minutes (70 minutes per week). At the end of each week, they will complete a brief survey to assess changes in treatment, and provide assessments of psychosocial wellbeing. At the end of the 8-week intervention period, participants will be emailed an online survey and be asked to complete a second blood draw, and compensation will be provided. At this time, participants will no longer be required to wear the sleep device, complete sleep diaries, or use their wellness app.

Participants then wait until the beginning of study week 20 to begin the follow-up period. At Week 20, for a period of 7 days, participants will be asked to wear the sleep device continuously and complete an online sleep diary each morning. They will also be asked to complete an online survey and provide a third blood sample. At the end of the follow-up week, participants will return their sleep device and receive their earned compensation.

ELIGIBILITY:
Inclusion Criteria:

1. Self-declared diagnosis of hematological cancer on stable maintenance management* by treating physician (i.e., on stable medical therapy) or observation (i.e., no changes in disease targeted medications for the past two weeks)
2. Not currently participating in a therapeutic pharmacologic clinical trial
3. Not planning to receive an allogenic stem cell transplantation during the study time frame (i.e., 20 weeks)
4. Score of >5 on PSQI (Pittsburgh Sleep Quality Index)
5. Own a mobile smartphone (iPhone with iOS 14 or later or an Android 6 or later) with an active data or WiFi connection
6. Willing to download two mobile apps
7. Able to read/understand English
8. ≥18 years of age
9. Willing to be randomized
10. Willing to drive to a nearby lab for blood draws 3x during the study over the course of 20 weeks (8-week intervention period followed by 12-week follow-up period)
11. Taking sleep medications and/or over-the-counter sleep drugs/supplements (if any) on fewer than 3 nights per week and one of the following: 1) willing to maintain the same intake without change throughout the study time frame (i.e., 20 weeks) or 2) willing to discontinue if intake is prescribed "as needed" (PRN) by a physician throughout the study time frame (i.e., 20 weeks)

Exclusion Criteria:

1. Self-report meditation practice or meditative movement practice (i.e., yoga, tai chi, qi gong) of ≥60 min/week in past 2 months
2. Reside outside of the United States of America
3. Any planned change to a new pharmacologic therapy (i.e., new drug) for the treatment of their cancer diagnosis (excluding dose changes)
4. Diagnosed with a sleep disorder except insomnia (≥2 positive categories on Berlin Questionnaire)
5. Taking prescribed sleep medications and/or over-the-counter drugs/supplements (including drugs like NyQuil, Benadryl, and other antihistamine-based drugs) on ≥3 nights per week
6. Any other diagnosed and uncontrolled medical or psychiatric condition
7. Has a pacemaker
8. Shift work schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sleep Disturbance (subjective) | Changes in sleep disturbance will be measured at baseline, week 2, week 4, week 6, week 8, and week 20. Total scores range from 0 to 28 with scores 8 to 14, and ≥15 indicating subclinical and moderate-to-severe insomnia symptom severity, respectively.
  Sleep disturbance will be measured with the Insomnia Severity Index (ISI). Total scores range from 0 to 28 with scores 8 to 14, and ≥15 indicating subclinical and moderate-to-severe insomnia symptom severity, respectively.
Sleep Disturbance (subjective) | Changes in sleep disturbance will be measured at baseline, week 8, and week 20. This form consists of 8 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
  Sleep disturbance will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8b. This form consists of 8 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
Sleep Disturbance (subjective) | Changes in sleep disturbance will be measured at baseline, week 8, and week 20. This form consists of 8 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
  Sleep disturbance will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment. This form consists of 8 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
Sleep disturbance (subjective) | Changes in sleep disturbance will be measured weekly throughout the 8-week intervention period and once again during the week 20 follow-up period.
  Sleep disturbance will be measured with an investigator-developed weekly sleep diary
Sleep disturbance (objective) | Changes in sleep disturbance will be measured weekly throughout the 8-week intervention period and once again during the week 20 follow-up period.
  Sleep disturbance will be measured with wrist actigraphy

SECONDARY OUTCOMES:
Inflammation | Changes in inflammation will be measured at baseline, week 8, and week 20.
  Inflammation will be measured with blood serum cytokines (C-reactive protein, TNF-a, IL-6, IL-8)
Fatigue (subjective) | Changes in fatigue will be measured at baseline, week 8, and week 20.
  Fatigue will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Adult Cancer Fatigue Short Form 7a. This form consists of 7 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
Anxiety (subjective) | Changes in anxiety will be measured at baseline, week 8, and week 20.
  Fatigue will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short Form 7a. This form consists of 7 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.
Depression (subjective) | Changes in fatigue will be measured at baseline, week 8, and week 20.
  Fatigue will be measured with the Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression Short Form 8a. This form consists of 8 items in a 1-5 Likert scale. The measure generates a total summed score, which is then converted to a standardized t-score.

OTHER OUTCOMES:
Wellness app engagement | Changes in engagement will be measured by minutes used per day/week on a weekly basis throughout the 8-week intervention period.
  Engagement with the wellness app will be tracked by user statistics

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — UT Health San Antonio
Locations (3):
- United States (3):
  - Arizona State University, Phoenix, Arizona
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Mays Cancer Center at The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huberty J, Bhuiyan N, Eckert R, Larkey L, Petrov M, Todd M, Mesa R. Insomnia as an Unmet Need in Patients With Chronic Hematological Cancer: Protocol for a Randomized Controlled Trial Evaluating a Consumer-Based Meditation App for Treatment of Sleep Disturbance. JMIR Res Protoc. 2022 Jul 1;11(7):e39007. doi: 10.2196/39007. PMID 35776489